CLINICAL TRIAL: NCT05036746
Title: Do Health Complaints in Adolescence Increase the Risk of Future Persistent Musculoskeletal Pain? Analyses From the Population-based Fit Futures Study
Brief Title: Health Complaints in Adolescence and Future Persistent Musculoskeletal Pain
Status: Completed | Type: Observational
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Britt Elin Øiestad, Professor, Oslo Metropolitan University
Other Study IDs: 2019/599B
Record Dates: First submitted 2021-09-02; First posted 2021-09-08 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Musculoskeletal Pain
Keywords: Musculoskeletal pain; Health complaints; Risk
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Persistent musculoskeletal (MSK) pain in adolescence is associated with disability, absence from school and reduced quality of life. We know little about risk factors and underlying mechanisms of persistent MSK pain in this age group. For example, the effect of other health complaints on the development of persistent MSK pain is scarcely investigated. In this prospective cohort study, data from the Fit Futures study on Norwegian adolescents (15-19 years old) will be used to investigate whether health complaints and an accumulation of health complaints in adolescence are associated with the incidence of persistent MSK pain two years later.

DETAILED DESCRIPTION:
There is a need of knowledge on risk factors and underlying mechanisms of persistent MSK pain in adolescence to increase our understanding and facilitate preventative strategies.

OBJECTIVE:

The aims of this prospective cohort study are to investigate whether health complaints and an accumulation of health complaints in adolescence, are associated with the incidence of persistent MSK pain two years later.

METHODS:

This will be a prospective study using data from the Fit Futures study conducted in the northern Norway. Adolescents (15-19 years) were recruited to the first survey (Fit Futures 1, FF1) in 2010/2011, and followed up to years later (Fit Futures 2, FF2). Data was collected through a comprehensive questionnaire and physical tests.

The exposures will be common health complaints in adolescence measured in FF1, including self-reported asthma, allergic rhinitis, atopic eczema, abdominal pain, headache and psychological distress (Hopkins Symptom Checklist).

Potential confounders will include age, sex and parents' socioeconomic status.

Statistical analyses:

Histograms and QQ-plots will be used to investigate the distribution of data. Normally distributed data will be presented with means and standard deviations (SD), while median and range will be used to present skewed data. Categorical data will be presented as counts and percentages. Missing data in exposures and confounders will be considered handled with multiple imputation. Participants with missing data on outcome will be excluded from the analyses. Baseline characteristics of adolescents lost to follow-up or with incomplete outcome data in FF2 will be compared to baseline characteristics of respondents.

A two-year incidence rate of persistent MSK pain will be presented.

Logistic regression analyses, providing odds ratios (ORs) with 95% confidence intervals (CI), will be used to investigate the association between health complaints (measured in FF1) and later persistent MSK pain (measured in FF2). The association between health complaints and persistent MSK pain will first be investigated separately for each complaint (asthma, allergic rhinitis, atopic eczema, psychological distress, headache and abdominal pain), secondly as the number of health complaints regardless of type (using an ordinal count variable). All logistic regression analyses will be conducted as crude and adjusted analyses. Statistical analyses will be conducted with STATA statistical software system.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents, 15-19 years old, participating in Fit Futures 1

Exclusion Criteria:

* Age > 19 years at baseline
* Adolescents reporting persistent musculoskeletal pain at baseline

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Norwegian adolescents, 15-19 years old
Sampling Method: Probability Sample
Enrollment: 1038 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2013-06-01 (Actual)

PRIMARY OUTCOMES:
Persistent musculoskeletal pain | Two years
  Persistent musculoskeletal pain was measured at the 2-year follow-up by the questions: "Do you have persistent or constantly recurring pain that has lasted for three months or more?", "if you have persistent and constantly recurring pain that has lasted for 3 months or more, how often do you have this pain?" and "if you have persistent or constantly recurring pain that has lasted for 3 months or more, where does it hurt?". Persistent musculoskeletal pain will in this study be defined as pain that persist or constantly recur on a weekly basis or more often, for minimum three months, in one or more of the following pain sites; neck, jaw/temporormandibular joint, upper back, lower back, chest, shoulder, arm/elbow, hand, hip, thigh/knee/shin, ankle/foot.

IPD SHARING:
Plan to Share IPD: No